CLINICAL TRIAL: NCT06001424
Title: Effect of Life Kinetik Training on Lower Limb Coordination in Ataxic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, heba ahmed khalifa, Ass. Prof. Dr. of Physical therapy for Neurology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/001987
Record Dates: First submitted 2021-01-17; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Multiple Sclerosis; Ataxia
Keywords: Multiple Sclerosis; ataxia; coordination; life kinetic exercises
MeSH Terms: conditions — Multiple Sclerosis; Ataxia | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: randomized controlled trail
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): will receive physical therapy program of in addition to life kinetik training.
  Interventions: Other: physical therapy; Other: life kinetic exercises
- control (Active Comparator): will receive physical therapy program
  Interventions: Other: physical therapy

INTERVENTIONS:
Other: physical therapy — Frenkel's exercises for lower limb, Proprioceptive neuromuscular facilitation for upper limb in the form of rhythmic stabilization
Other: life kinetic exercises — A multimodal training that combines coordinative, cognitive and visual tasks.
  Arms: study group

SUMMARY:
Coordination is essential for the performance of most daily motor activities. Coordination problems are common in MS patients. One of the most commonly reported symptoms is dysmetria (limb ataxia). Ataxia is thought to occur in about 80% of MS patients. It leads to limitations in daily life activities. Aim of Study: to investigate the effect of life kinetik training on lower limb coordination in MS patients with ataxia.

DETAILED DESCRIPTION:
Methods: Thirty remitting relapsing Multiple Sclerosis (RRMS) patients from both sexes with ataxic symptoms, will be recruited from multiple sclerosis specialized clinic in the Neurology department, Faculty of Medicine, Cairo University with EDSS score will be ranged from 2 to 4 and SARA score will be ranged from 1 to 10. Lower Extremity Motor Coordination Test (LEMOCOT) will be used to assess lower limb motor coordination. They will be randomly assigned into two equal groups; control group (GI) will receive selected physical therapy program and study group (GII) will receive same program of (GI) in addition to life kinetik training.

ELIGIBILITY:
Inclusion Criteria:

* MS from both sexes
* Patients' age will be ranged from 20 to 45 years
* Expanded disability scale (EDSS) score ranging from "two" to "four"

Exclusion Criteria:

* Patients with Ataxia caused by other cause rather than MS
* Patients with other neurological disease or orthopedic deformities may affect movement
* Patients with cardiovascular and pulmonary diseases that make exercise unsafe
* Patients with cognitive impairment or psychiatric disorders

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-24 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-29 (Actual)

PRIMARY OUTCOMES:
Lower Extremity Motor Coordination Test (LEMOCOT) | at baseline
  test to assess lower limb coordination
Lower Extremity Motor Coordination Test (LEMOCOT) | post intervention (after one month)
  test to assess lower limb coordination

SECONDARY OUTCOMES:
Four Square Step Test (FSST) | at baseline
  test to assess dynamic balance
Four Square Step Test (FSST) | post intervention (after one month)
  test to assess dynamic balance

CONTACTS AND LOCATIONS:
Overall Officials: Moshera H Darwish, Prf. Dr, Study Director — Professor of Physical therapy for Neurology
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edwards EM, Fritz NE, Therrien AS. Cerebellar Dysfunction in Multiple Sclerosis: Considerations for Research and Rehabilitation Therapy. Neurorehabil Neural Repair. 2022 Feb;36(2):103-106. doi: 10.1177/15459683211065442. Epub 2021 Dec 21. PMID 34931569